CLINICAL TRIAL: NCT05729503
Title: SPG Block Versus Placebo to Manage Anxiety at Electronic Dance Music Festivals
Brief Title: Effect of SPG Block for Patients With Anxiety at Electronic Dance Music Festivals
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REB23-0181
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2% Lidocaine (Experimental): 1 cotton tip applicator, pre-soaked in 2% lidocaine, inserted into each nare, and left for 10 minutes
  Interventions: Drug: Lidocaine 2% Injectable Solution
- Placebo (Placebo Comparator): 1 cotton tip applicator, pre-soaked in saline, inserted into each nare, and left for 10 minutes
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine 2% Injectable Solution — Cotton tip applicator pre-soaked with lidocaine
  Other Names: Lidocaine
  Arms: 2% Lidocaine
Drug: Placebo — Cotton tip applicator pre-soaked with saline
  Other Names: Saline
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn about the effect of a sphenopalatine ganglion (SPG) block in anxious patients at electronic dance music festivals. The main question is:

- Is an SPG block useful in reducing anxiety, in comparison to placebo?

Participants will have lidocaine-soaked cotton tip applicator placed inside each nare for 10-minutes, or have a saline-soaked cotton tip applicator placed inside each nare for 10-minutes.

Researchers compare the lidocaine-soaked intervention (SPG block) with the saline-soaked intervention (placebo) to see if it reduces anxiety in patients presenting at electronic dance music festivals with anxiety.

DETAILED DESCRIPTION:
1. Background & Rationale

   Electronic dance music festivals are a growing source of entertainment in Canada. Attended by thousands at a time, it is important to have a medical team onsite to manage clinical issues in these mass gatherings. One of the most common clinical presentations at these festivals is anxiety. In a low-resource setting, it is not always possible to supply all guests with oral or injectable anti-anxiety therapy. Additionally, anti-anxiety medication is often sedating, which we would want to avoid in a patient population at higher risk of sedation (e.g., intoxication). A simple, non-sedating, alternative treatment that can be administered by a medical team member that can be given without the need of a needle would be ideal.

   Anecdotal reports have noted that sphenopalatine ganglion (SPG) blocks with lidocaine, intranasally, is effective for the relief of anxiety. As well, the PI has had anecdotal success in managing patient anxiety with SPG blocks. At the time of writing, there has been no published study found by our team to evaluate the efficacy of SPG blocks on anxiety.
2. Research Question & Objectives

   Question: In electronic dance music festival attendees, who present with anxiety to the medical team, how does a 2% lidocaine-soaked cotton tip applicator, inserted into both nares until it meets resistance, compare with a saline-soaked cotton tip applicator, inserted into both nares until it meets resistance, for self-reported anxiety 10-minutes post-intervention?

   The objective of this trial is to study the effectiveness of bilateral SPG block for anxiety.
3. Methods

All individuals, who present with anxiety to the main medical area at electronic dance music festivals in Canada, will be recruited until sample size reaches at least 70 people. Inclusion criteria will include festival attendees aged 18+ with a complaint of anxiety. Exclusion criteria will include known allergy to lidocaine (standard practice involves medical team members asking patients what allergies they have), inability to pass a cotton tip applicator through the nares (e.g., obstruction), inability to report level of anxiety, or already have taken an anti-anxiety medication (e.g., lorazepam, midazolam).

After obtaining consent, participants will be randomized into two study arms using a random number generator. Arm 1 will receive an intranasal SPG block with 2% lidocaine in each nare, applied with long cotton tip applicators. Arm 2 will receive a long cotton tip applicator soaked with saline, inserted in each nare (placebo). The cotton tip applicators will remain in the nares for 10 minutes before removal.

After randomization, participants will be asked to rate their anxiety on a numeric response scale (0 to 10, where 0 is no anxiety and 10 is "worst anxiety imaginable") prior to receiving their assigned intervention. 10-minutes following intervention, participants will be asked to rate their anxiety once more.

ELIGIBILITY:
Inclusion Criteria:

* Festival attendees aged 18+
* A complaint of anxiety of at least 1 on a scale of 0 to 10 (11-point scale, where 0 represents "no anxiety" and 10 represents "worst anxiety imaginable").

Exclusion Criteria:

* Known allergy to lidocaine (standard practice involves medical team members asking patients what allergies they have; we will not directly ask about lidocaine in order to keep participants blinded to interventions)
* Inability to insert cotton tip applicator through the nares (e.g., distorted nasal anatomy, active nosebleed, obstructed nasal passages)
* Inability to verbally report level of anxiety
* Prior administration of an oral or intravenous anti-anxiety medication (e.g., lorazepam, midazolam) by festival medical staff since arrival at the festival (would confound treatment effect)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-05-06 (Estimated); Primary Completion 2026-05-06 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Patients' self-reported anxiety scores post-intervention | 10-minutes post-intervention
  Patients will rate their anxiety on an 11-point scale (0 = "no anxiety", 10 = "worst anxiety imaginable"). The lowest score is 0 and the highest score is 10. Lower scores indicate better outcome.

SECONDARY OUTCOMES:
Use of rescue-medication (i.e., oral/intravenous anti-anxiety medication) | 10-minutes post-intervention
  Presence (1) or absence (0) of any rescue-medication, (i.e. oral/intravenous anti-anxiety medication), identified by patient's chart
Improvement of headache | 10-minutes post-intervention
  Yes, No, or N/A. For patients who had a headache prior to the intervention, these patients will answer whether the intervention improved their headache. This is because it is known that SPG blocks improve headaches. There is a possibility that anxiety may be improved, because a headache is improved.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony V Seto, MD, Principal Investigator — University of Calgary
Locations (4):
- Canada (4):
  - Electronic Dance Music festivals in Calgary, Calgary
  - Electronic Dance Music festivals in Edmonton, Edmonton
  - Electronic Dance Music festivals in Toronto, Toronto
  - Electronic Dance Music festivals in Vancouver, Vancouver

IPD SHARING:
Plan to Share IPD: No